CLINICAL TRIAL: NCT06190860
Title: Platelet Rich Fibrin as a Modulator of the Wound Healing Response in Smokers
Brief Title: Platelet Rich Fibrin Treatment for the Alveolar Ridge Preservation in Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1181007
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Alveolar Process Atrophy; Smoking, Cigarette; Platelet-Rich Fibrin
MeSH Terms: conditions — Alveolar Bone Loss; Cigarette Smoking | interventions — Biopsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Post-extraction sockets will be sutured and left to heal spontaneously with physiological blood clot.
  First intervention: intraoral scan and intraoral scan and Cone Beam Computed Tomography in the treated zone. Clinicians will make a post-surgical control to evaluate how healing will be performed Four months after the first Intervention, participants will recall getting a second scan and Cone Beam Computed Tomography in the treated zone. Images will be used for implant treatment planification. Before implant placement, a biopsy (2 mm in diameter) will be taken. The biopsy will be analyzed by Micro-computed tomography and decalcified and included in paraffin for histological sections.
  Interventions: Other: Intraoral Scan; Radiation: Computed Tomography; Other: Biopsy
- L-PRF Treatment (Experimental): Post-extraction sockets will be treated with L-PRF plugs and membranes. First intervention: intraoral scan and intraoral scan and Cone Beam Computed Tomography in the treated zone. Clinicians will make a post-surgical control to evaluate how healing will be performed Four months after the first Intervention, participants will recall getting a second scan and Cone Beam Computed Tomography in the treated zone. Images will be used for implant treatment planification. Before implant placement, a biopsy (2 mm in diameter) will be taken. The biopsy will be analyzed by Micro-computed tomography and decalcified and included in paraffin for histological sections.
  Interventions: Other: Autologous Leukocyte and platelet-rich fibrin; Other: Intraoral Scan; Radiation: Computed Tomography; Other: Biopsy

INTERVENTIONS:
Other: Autologous Leukocyte and platelet-rich fibrin — Participants will be treated with L-PRF plugs and membranes from autologous venous blood. Participants will have drawn blood after venipuncture (median cubital vein) into sterile, glass-coated plastic 9 mL tubes without anticoagulant. These tubes will be centrifuged at 2700 rpm for 12 min (Relative Centrifugal Forces-clot = 408 g). After tooth extraction, participants in the experimental group will be treated with L-PRF plugs and membranes.
  Arms: L-PRF Treatment
Other: Intraoral Scan — Intraoral scan will be taken in the treated zone after tooth extraction and after four months.
Radiation: Computed Tomography — Cone Beam Computed Tomography in the treated zone will be taken after tooth extraction and after four months.
Other: Biopsy — Before dental implant placement, a biopsy (2 mm in diameter) will be taken. The biopsy will be analyzed by Micro-computed tomography and decalcified and included in paraffin for histological sections.

SUMMARY:
Bone healing is affected by smoking, particularly healing of extraction sockets, showing deficiencies in vertical and horizontal bone dimensions compared to the healing of non-smokers. Several approaches have been made to stimulate.

Bone wound healing, including human autologous blood-derived fractions. One of these fractions is the leukocyte platelet-rich fibrin (L-PRF).

L-PRF has been evidenced as potentially beneficial in promoting bone defect filling in alveolar bone and socket preservation in non-smokers. However, scarce evidence is related to this beneficial effect in smokers.

This clinical trial aims to study and compare the in vivo effects of L-PRF during bone wound healing and regeneration in smokers.

The main question is:

Has the L-PRF a beneficial effect during alveolar ridge preservation in smokers? After consent, participants with tooth extraction indications and implant rehabilitation treatment will be enrolled. After randomization, participants will be assigned to an experimental group treated with L-PRF plugs and membranes or a control group (physiological healing).

Participants will receive two interventions:

* First intervention: Tooth extraction, intraoral scan, and Cone Beam Computed Tomography in the treated zone.
* Second intervention (4 months after first intervention): intraoral scan and Cone Beam Computed Tomography in the treated zone

DETAILED DESCRIPTION:
* This study will be conducted according to the principles outlined in the Declaration of Helsinki regarding experiments on human beings. This work was submitted and approved by the Ethics and Scientific Committee, approval number ID170706007.
* Participant selection: Volunteers must agree to participate in the study after signing an informed consent (previously approved by the Ethics Committee). Participants will be treated at the Dental Clinical School of Dentistry at the Pontificia Universidad Católica de Chile or in the Dentistry/ Health Sciences Center at San Bernardo from the University of the Andes, Chile. Both institutions are located in Santiago, Chile.

Diagnosis and evaluation before interventions: Volunteer participants will be selected after a clinical and periapical radiographic examination to establish the need for tooth extraction. Laboratory tests, including a complete blood coagulation profile, will be required for all volunteers. Finally, a salivary cotinine test will ensure the smoker's condition.

* Randomization: A random number will be assigned to all participants. An independent research team member will establish a randomization sequence without contact with the clinician's team. Sealed envelopes with randomization will be performed and opened by surgeons before the tooth extraction.
* First Intervention: Participants assigned to the experimental group will be treated with L-PRF plugs and membranes from venous blood. Participants will have drawn blood after venipuncture (median cubital vein) into sterile, glass-coated plastic 9 mL tubes without anticoagulant. These tubes will be centrifuged at 2700 rpm for 12 min (Relative Centrifugal Forces-clot = 408 g). After tooth extraction, participants in the experimental group will be treated with L-PRF plugs and membranes, and the control group will be sutured. Participants in both groups will be intraoral scan and intraoral scan and Cone Beam Computed Tomography in the treated zone. Clinicians will make a post-surgical control to evaluate how healing will be performed.
* Second Intervention: Four months after the first Intervention, participants will recall getting a second scan and Cone Beam Computed Tomography in the treated zone. Images will be used for implant treatment planification. Before implant placement, a biopsy (2 mm in diameter) will be taken. The biopsy will be analyzed by Micro-computed tomography and decalcified and included in paraffin for histological sections.
* The primary outcome variable established will be radiographic linear changes in horizontal width and vertical height of the alveolar ridge measured in the CBCTs taken immediately after tooth extraction and after four months. Secondary outcomes included the changes in ridge contours and volume estimated from the intraoral scan images.
* Data analysis: Members of the research team who do not know the group intervention of the participants will determine alveolar ridge height and width in oral scans and CBCTs taken in the first and second Interventions. As such, micro-CT analysis and histological sections will be analyzed.
* Statistical analysis The results will express the mean ± 95% CI. Will be considered as significant differences when P < 0.05. Nominal data will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Smokers (at least five cigarettes/day) have had the habit for at least one year.

* treatment plan that includes the indication of extraction of a single, double-rooted, or multi-rooted tooth and prosthetic rehabilitation with osseointegrated implants
* Patients with controlled systemic pathologies (hypertension, diabetes, hypercholesterolemia).
* With alveolar bone support of at least 50% and whose indication is delayed implant placement at least four months after extraction.
* Periapical lesions of no more than 5 mm diameter.

Exclusion Criteria:

* patients taking immunosuppressive or anticoagulant drugs
* pregnant
* users of removable prostheses
* Individuals with altered values of platelet count or coagulation parameters.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-05-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge changes | inmediately after tooth extraction and after four months
  linear changes in horizontal width and vertical height of the alveolar ridge measured in the CBCTs taken immediately after tooth extraction and after four months.

SECONDARY OUTCOMES:
Alveolar ridge sof tissue changes | inmediately after tooth extraction and after four months
  changes in ridge contours and volume estimated from the intraoral scan images
Tissue healing | Biopsy at least four months after tooth extraction
  Tissue analysis by Micro-CT and histological sections.

CONTACTS AND LOCATIONS:
Overall Officials: Constanza Martínez, DDS PhD, Principal Investigator — University of the Andes, Chile
Locations (2):
- Chile (2):
  - Clinical Facility, School of Dentistry, Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan
  - Dental facility, Health center at San Bernardo, Faculty of Dentistry, University of the Andes, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will underlie results in a publication.
Supporting Information: Study Protocol, CSR